CLINICAL TRIAL: NCT04630314
Title: Procedural and 1-year Outcomes Following Large Vessel Coronary Artery Perforation Treated by Covered Stents Implantation: Multicentre CRACK Registry
Brief Title: Covered Stents in Treatment of Coronary Artery Perforation
Acronym: CRACK
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Wojciech Wańha, MD, PhD, Medical University of Silesia
Other Study IDs: 04
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Coronary Artery Perforation
Keywords: Percutaneous coronary intervention; Coronary artery perforation; Covered stent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive patients treated with covered stents post PCI CAP
  Interventions: Device: Percutaneus Coronary Intervention

INTERVENTIONS:
Device: Percutaneus Coronary Intervention — Covered Stent

SUMMARY:
Covered stents have been mainly used for treatment of potentially life-threatening coronary artery perforation and coronary artery aneurysm. Prior studies suggest that the use of covered stents improves event-free survival, enabling a life-threatening situation to be managed without emergency surgery and with significantly reduced rates of mortality, cardiac tamponade, and major adverse cardiac events. Although the devices are used for a long time, very limited study has described procedural-related outcomes with this specific technology. We therefore want to report procedural, in-hospital and long term outcomes among patients treated with the covered stents.

ELIGIBILITY:
Inclusion Criteria:

* Iatrogenic, peri-PCI CAP treated with covered stent implantation

Exclusion Criteria:

* CAP caused due to other cause than PCI
* PCI of other vascular territories during the same procedure

Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 1 year
  MACE

SECONDARY OUTCOMES:
Stent Thrombosis (ST) | 1 year
  ST
Cardiac Death | 1 year
  CV Death
Target Lesion Revascularization (TLR) | 1 year
  TLR
Myocardial Infarction (MI) | 1 year
  MI

CONTACTS AND LOCATIONS:
Locations (6):
- Poland (6):
  - Department of Invasive Cardiology, Medical University of Białystok, Bialystok
  - First Department of Cardiology, Medical University of Gdansk, Gdansk
  - Wojciech Wańha, Katowice
  - Second Department of Cardiology, Jagiellonian University Medical College, Krakow
  - Miedziowe Centrum Zdrowia S.A., Lubin
  - Third Department of Cardiology, Medical University of Katowice, Zabrze